CLINICAL TRIAL: NCT02769442
Title: Prospective, Randomized Controlled Comparison of TERUMO SurFlash Plus Versus BD Insyte Autoguard in an Urban ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Principal Investigator, Siamak Moayedi, MD, PI, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00068278
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Catheters; Catheterization, Peripheral
Keywords: Intravenous; Catheter; Puncture; Peripheral Catheterization; First Stick Success; Contamination; Terumo; SurFlash
MeSH Terms: interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terumo SurFlash Plus catheter (Experimental): Patients randomized to the Terumo catheter
  Interventions: Device: Terumo SurFlash Plus catheter
- BD Insyte Autoguard catheter (Active Comparator): Patients randomized to the BD catheter
  Interventions: Device: BD Insyte Autoguard catheter

INTERVENTIONS:
Device: Terumo SurFlash Plus catheter
  Arms: Terumo SurFlash Plus catheter
Device: BD Insyte Autoguard catheter
  Arms: BD Insyte Autoguard catheter

SUMMARY:
A randomized prospective comparison of two FDA approved intravenous catheters in the emergency department setting. The Terumo SurFlash Plus offers novel technologies that promise to increase intravenous access success rates and decrease blood contamination of the insertion site. This study would analyze these properties in our busy, urban emergency department setting where time and safety of intravenous access are most critical.

DETAILED DESCRIPTION:
Rational for the Study Emergency department (ED) patients frequently require rapid, short-term intravenous (IV) access for diagnosis and treatment of emergency medical conditions. IV access can be uncomfortable and painful for the patient. Therefore ensuring first attempt success is important. Furthermore, given the time-sensitive nature of emergent medical conditions, immediate success helps to minimize delay in analgesic medication administration, resuscitation and therapeutic interventions. The process of obtaining IV access has the potential for operator exposure to blood-borne pathogens. After a tourniquet is placed on an extremity, positive venous pressure forces blood out of the catheter until a lure lock can be applied. Traditional IV catheters require the operator to kink the catheter and apply pressure to the body of the catheter to mitigate the degree of blood leakage while simultaneously connecting the lure lock. This is a complicated process that often leads to blood contamination of the insertion site, and the environment, including the potential for blood spillage on the bedding, ground or the operator. In addition to the potential for blood-born pathogen exposures, this spillage leads to further patient care delays, as it requires prompt cleaning.

Terumo Medical Corp., a leading manufacturer of medical devices, has introduced a novel IV access catheter (which is already FDA approved) with features that promise to increase first attempt success and decrease blood contamination during the insertion process. The Terumo SurFlash Plus catheter has a technology that produces a visible flash of blood at the end of the catheter when the needle is placed in the vessel and a second flash between the catheter and the needle which confirms proper catheter placement in the vein. Furthermore, this new catheter has a proprietary safety valve that minimizes the risk of blood exposure between needle removal and IV lure lock attachment.

This study would analyze these unique properties (first skin puncture success and insertion site blood contamination) in a high volume, urban emergency department where time and safety of IV access are critical.

Purpose of Study Primary Objective: Compare the rate of first-skin puncture success using the Terumo SurFlash Plus compared with the BD Insyte Autoguard.

Secondary Objective: Compare the frequency and severity of blood contamination of the insertion site between the two aforementioned devices.

Research Design This will be a prospective, randomized controlled study of the Terumo SurFlash Plus IV catheter versus the current standard ED IV catheter (BD Insyte Autoguard).

Study device: The Terumo SurFlash Plus catheter is FDA approved and already used at multiple medical centers in the United States. Gauge sizes 18, 20 and 22 will be provided by TERUMO to the ED at no cost to the hospital.

IV inserters (operators) will be Mercy Medical Center emergency department technicians, nurses and providers who routinely obtain IV access in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Adult ED patient requiring an IV for clinical care
* Hemodynamically stable: pulse >50 and <130, MAP>60
* Willing to read (or be read to) the informed consent and participate in study

Exclusion Criteria:

* Medically unstable
* Agitated or psychiatrically unstable
* Lacking capacity to consent, such as with altered mental status.
* Unable to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Moayedi, MD, Principal Investigator — Assistant Professor
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Youtube video describing Terumo SurFlash Plus catheter — https://www.youtube.com/watch?v=5ww5tgnPuXg

RESULTS

PARTICIPANT FLOW:
Groups:
- Becton Dickinson (BD) Insyte Autoguard Catheter: Patients randomized to the Becton Dickinson (BD) catheter
Period: Overall Study
Arm/Group | Terumo SurFlash Plus Catheter | Becton Dickinson (BD) Insyte Autoguard Catheter
Started | 309 | 291
Completed | 309 | 291
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terumo SurFlash Plus Catheter | BD Insyte Autoguard Catheter | Total
Number analyzed (Participants) | 309 | 291 | 600
Age, Customized [Mean (Standard Deviation); unit: years]
  Patient Age Mean | 51.1 (17.7) | 50.9 (17.7) | 51 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 175 | 376
  Male | 108 | 116 | 224
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First-skin Puncture Success
Description: 1. First attempt success, defined as one skin puncture (redirection permitted) which allows for completion of a blood draw and/or flush without extravasation.
  2. Gauge size
  3. Patient prior history of difficult IV access
  4. Operator type (ED Technician/Registered Nurse/Physician Assistant/Nurse Practitioner/Resident/Attending)
  5. Operator years of experience with IV access
  6. Type of catheter used
Time Frame: Within first minute of IV access
Measure: Count of Participants; unit: Participants
Arm/Group | Terumo SurFlash Plus Catheter | BD Insyte Autoguard Catheter
Number analyzed (Participants) | 309 | 291
Participants | 244 | 229

2. Secondary Outcome: Number of Participants With Blood Visible at Site of Insertion
Description: Compare the frequency of bleeding near the insertion site
Time Frame: Within first minute of IV access
Measure: Number; unit: participants
Arm/Group | Terumo SurFlash Plus Catheter | BD Insyte Autoguard Catheter
Number analyzed (Participants) | 309 | 291
participants | 8 | 92

ADVERSE EVENTS:
Time Frame: 6 hours or less depending on duration of emergency department stay
Arm/Group | Terumo SurFlash Plus Catheter | BD Insyte Autoguard Catheter
All-Cause Mortality (participants affected / at risk) | 0/309 | 0/291
Serious Adverse Events (participants affected / at risk) | 0/309 | 0/291
Other Adverse Events (participants affected / at risk) | 0/309 | 0/291

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No